CLINICAL TRIAL: NCT05840159
Title: A Phase 4 Study of a 3-Day vs. 7-Day Regimen of Doxycycline for the Treatment of Chlamydial Infection
Brief Title: A Study of Doxycycline to Treat Chlamydial Infection
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-0019; 5UM1AI148684-03 (NIH)
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-04-22

CONDITIONS: Chlamydial Infection
Keywords: Chlamydia; Doxycycline; Infection; intervention; Phase 4
MeSH Terms: conditions — Chlamydia Infections; Infections | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm 1 (Experimental): 100 mg of doxycycline orally administered twice daily for 3 days and 4 days of placebo to assigned women participants >/= 16 years old with confirmed urogenital Chlamydia trachomatis (CT). N=166.
  Interventions: Drug: Doxycycline; Other: Placebo
- Arm 2 (Active Comparator): 100 mg of doxycycline orally administered twice daily for 7 days to assigned women participants >/= 16 years old with confirmed urogenital Chlamydia trachomatis (CT). N=166.
  Interventions: Drug: Doxycycline
- Arm 3 (Experimental): 100 mg of doxycycline orally administered twice daily for 3 and 4 days of placebo days to assigned men participants >/= 16 years old with confirmed rectal Chlamydia trachomatis (CT). N=166.
  Interventions: Drug: Doxycycline; Other: Placebo
- Arm 4 (Active Comparator): 100 mg of doxycycline orally administered twice daily for 7 days to assigned men participants >/= 16 years old with confirmed rectal Chlamydia trachomatis (CT). N=166.
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — Doxycycline is a synthetic tetracycline derivative with similar antimicrobial activity.
Other: Placebo — Placebo
  Arms: Arm 1; Arm 3

SUMMARY:
This is a Phase 4 blinded, randomized, active-controlled, non-inferiority trial. Final evaluable population will include a minimum 596 individuals: 298 women with confirmed urogenital chlamydia (CT) and 298 men with confirmed rectal chlamydia (CT). Approximately 664 participants will be enrolled to achieve a minimum 596 participants who contribute primary outcome data. Randomization will be stratified by study site and sex: 332 women and 332 men. Participants will be randomized 1:1 to a 3-day regimen of doxycycline or a 7-day regimen of doxycycline. The study blind will be maintained by providing 7 days of identical pre-filled blister packs, one with 3 days of active treatment and 4 days of placebo, and the other with 7 days of active treatment. Participants will be asked to return 28 days after randomization (at day 29), at which time they will be re-tested for chlamydia (CT) using a laboratory-based chlamydia (CT) nucleic acid amplification test (NAAT).

DETAILED DESCRIPTION:
This is a Phase 4 blinded, randomized, active-controlled, non-inferiority trial. Final evaluable population will include a minimum 596 individuals: 298 women with confirmed urogenital chlamydia (CT) and 298 men with confirmed rectal chlamydia (CT). Approximately 664 participants will be enrolled to achieve a minimum 596 participants who contribute primary outcome data. Randomization will be stratified by study site and sex: 332 women and 332 men. Participants will be randomized 1:1 to a 3-day regimen of doxycycline or a 7-day regimen of doxycycline. The study blind will be maintained by providing 7 days of identical pre-filled blister packs, one with 3 days of active treatment and 4 days of placebo, and the other with 7 days of active treatment. Participants will be asked to return 28 days after randomization (at day 29), at which time they will be re-tested for chlamydia (CT) using a laboratory-based chlamydia (CT) nucleic acid amplification test (NAAT).

The primary objective is to compare the efficacy of a 3-day vs. 7-day regimen of doxycycline for treatment of urogenital chlamydia (CT) infection in women based on proportion of participants with microbiologic cure (negative nucleic acid amplification test [NAAT] of vaginal swab and no positive nucleic acid amplification test (NAAT) of vaginal swab between study treatment and Day 29) at Day 29. Also, to compare the efficacy of a 3-day vs. 7-day regimen of doxycycline for treatment of rectal chlamydia (CT) infection in men based on proportion of participants with microbiologic cure (negative nucleic acid amplification test (NAAT) of rectal swab and no positive nucleic acid amplification test (NAAT) of rectal swab between study treatment and Day 29) at Day 29. The secondary objectives are to compare the efficacy of a 3-day vs. 7-day regimen of doxycycline for treatment of rectal CT infection in women based on microbiologic cure. Also, to compare the efficacy of a 3-day vs. 7-day regimen of doxycycline for treatment of urethral CT infection in men based on microbiologic cure. In addition, compare the efficacy of a 3-day vs. 7-day regimen of doxycycline for treatment of total CT infection (any anatomic site) in women and men based on microbiologic cure. Lastly, to compare the efficacy of a 3-day vs. 7-day regimen of doxycycline for treatment of rectal CT infection in men based on microbiologic cure, stratified by lymphogranuloma venereum (LGV) status.

ELIGIBILITY:
Inclusion Criteria:

1. Has untreated urogenital chlamydia (CT) (in women) or rectal CT (in men), diagnosed with a positive nucleic acid amplification test (NAAT) (point-of care or laboratory-based)* result within 14 days

   *Point-of-care (POC) test may or may not be FDA-cleared for CLIA waiver for diagnosis depending upon anatomic site of infection.
2. Must be age >/=16 years (where the IRB permits individuals aged 16-17 years old to consent to research); otherwise age >/= 18 years
3. Willing and able to understand and provide written informed consent before initiation of any study procedures
4. Willing to complete a 7-day study drug regimen
5. Willing to abstain from condomless anal or vaginal sex during the trial
6. Willing and able to adhere to planned study procedures for all study visits
7. Has valid contact information

Exclusion Criteria:

1. For women: lower abdominal or pelvic pain or other signs or symptoms consistent with a clinical diagnosis of pelvic inflammatory disease (PID) Per the CDC's 2021 STD Treatment Guidelines or refer to local guidelines.
2. Signs and symptoms that, in the judgement of a qualified clinician, warrant a prolonged course of treatment with doxycycline For example, 21 days of doxycycline for presumed lymphogranuloma venereum infection.
3. Received antimicrobial therapy active against C. trachomatis within 21 days prior to positive chlamydia (CT) test result, or between the positive chlamydia (CT) test result and study enrollment Use of the following antibiotics is exclusionary: doxycycline and related tetra- or glycylcyclines, macrolides (including azithromycin), fluoroquinolones, rifampin, quinupristin-dalfopristin, and linezolid. Note: Amoxicillin, penicillin, ceftriaxone, and other beta-lactam antibiotics are not considered exclusionary for this study.
4. Planning to take antimicrobial therapy active against chlamydia (CT) during the study period (e.g. doxycycline post-exposure prophylaxis, treatment for Mycoplasma genitalium infection, acne, or any other non-STI medical condition).
5. Currently enrolled in or plan to enroll in another study using antimicrobial therapy active against C. trachomatis during the study period
6. Pregnant or lactating, or plan to become pregnant within the study period
7. Known moderate to severe allergy to tetracyclines, excluding tetracycline-induced photosensitivity.
8. Plan to move or travel to another location that would preclude study follow-up appointments in clinic in the next 30 days
9. Use of a medication contraindicated to treatment with doxycycline within 7 days prior to enrollment or during the study period (systemic retinoids, barbiturates, carbamazepine, phenytoin, warfarin)
10. Previous enrollment in this trial
11. Any condition that, in the judgment of the investigator, precludes participation because it could affect participant safety or determination of study endpoints.

Of note, the following factors will NOT exclude participants from the study:

* Concomitant untreated gonorrhea (rectal, pharyngeal, or urethral) or known exposure to gonorrhea in the time between CT testing and study enrollment. Gonococcus (GC) infection identified during the course of pre-screening or screening will be treated per clinic standard practice and in accordance with local guidelines without concomitant azithromycin or other treatment for Chlamydia trachomatis infection.
* Clinical diagnosis of concomitant untreated primary or secondary syphilis or known exposure to syphilis
* Urethritis among men
* Contraception status
* Diagnosis of HIV

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of assigned men participants with microbiologic cure as detected via rectal swab | Day 1 through Day 29
  A participant with microbiologic cure is defined as having a negative Chlamydia trachomatis (CT) Nucleic Acid Amplification Test (NAAT) at Day 29 and no positive CT NAATs between study treatment and Day 29
Proportion of assigned women participants with microbiologic cure as detected via vaginal swab | Day1 through Day 29
  A participant with microbiologic cure is defined as having a negative Chlamydia trachomatis (CT) Nucleic Acid Amplification Test (NAAT) at Day 29 and no positive CT NAATs between study treatment and Day 29.

SECONDARY OUTCOMES:
Proportion of assigned men participants with microbiologic cure as detected via urine | Day 1 through Day 29
  A participant with microbiologic cure is defined as having a negative Chlamydia trachomatis (CT) Nucleic Acid Amplification Test (NAAT) at Day 29 and no positive CT NAATs between study treatment and Day 29.
Proportion of assigned men participants with microbiologic cure at all anatomic sites that were positive at baseline | Day 1 through Day 29
  A participant with microbiologic cure is defined as having a negative Chlamydia trachomatis (CT) Nucleic Acid Amplification Test (NAAT) at Day 29 and no positive CT NAATs between study treatment and Day 29.
Proportion of assigned women participants with microbiologic cure as detected via rectal swab | Day 1 through Day 29
  A participant with microbiologic cure is defined as having a negative Chlamydia trachomatis (CT) Nucleic Acid Amplification Test (NAAT) at Day 29 and no positive CT NAATs between study treatment and Day 29.
Proportion of assigned women participants with microbiologic cure at all anatomic sites that were positive at baseline | Day1 through Day 29
  A participant with microbiologic cure is defined as having a negative Chlamydia trachomatis (CT) Nucleic Acid Amplification Test (NAAT) at Day 29 and no positive CT NAATs between study treatment and Day 29.
Proportion of lymphogranuloma venereum (LGV)-negative assigned men participants with microbiologic cure as detected via rectal swab. | Day 1 through Day 29
  A participant with microbiologic cure is defined as having a negative Chlamydia trachomatis (CT) Nucleic Acid Amplification Test (NAAT) at Day 29 and no positive CT NAATs between study treatment and Day 29.
Proportion of lymphogranuloma venereum (LGV)-positive assigned men participants with microbiologic cure as detected via rectal swab. | Day 1 through Day 29
  A participant with microbiologic cure is defined as having a negative Chlamydia trachomatis (CT) Nucleic Acid Amplification Test (NAAT) at Day 29 and no positive CT NAATs between study treatment and Day 29.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - University of Alabama at Birmingham School of Medicine - Infectious Disease, Birmingham, Alabama
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown - Emory Clinic Infectious Diseases, Atlanta, Georgia
  - University of Rochester Medical Center - Vaccine Research Unit, Rochester, New York
  - University of Washington - Harborview Medical Center - Center for AIDS and STD, Seattle, Washington
- Kenya (2):
  - Pwani Research Centre, Mombasa
  - KEMRI-CCR PHRD Project, Thika

DOCUMENTS (1):
  • Informed Consent Form (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT05840159/ICF_000.pdf